CLINICAL TRIAL: NCT02614144
Title: Identifying Agents of Early-onset and Late-onset Nosocomial Pneumonia in Patients in Intensive Care Through Genetic Analysis of Bacterial DNA and Determination of Their Distribution.
Brief Title: Epidemiology of Hospital Acquired Pneumonia
Acronym: HAP
Status: Completed | Type: Observational
Sponsor: University Hospital Olomouc (Other)
Responsible Party: Principal Investigator, Radovan Uvizl, Radovan Uvizl, M.D., Ph.D., University Hospital Olomouc
Other Study IDs: IGA MZČR NT 14263-3/2013
Record Dates: First submitted 2015-11-20; First posted 2015-11-25 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Respiratory Tract Infection Bacterial
Keywords: Hospital Acquired Pneumonia; Mortality
MeSH Terms: conditions — Healthcare-Associated Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Biospecimen Retention: Samples With DNA — In intubated patients, secretion samples for microbiology culture tests are obtained by aspiration from the lower airway.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This project aimed at analyzing and assessing of the early and late Hospital-Acquired Pneumonia(HAP) bacterial pathogens and their resistance to antimicrobial agents. The incidence of their resistance to antimicrobial agent is assessed. Included are patients hospitalized in the Intensive Care Departments of cooperated University hospitals, who developed early or late HAP. Bacterial pathogens and their resistance to antibiotics are identified using standard microbiological methods. The patient's mortality with respect to their initial antibiotic therapy is statistically analyzed.

DETAILED DESCRIPTION:
Introduction. Hospital-acquired pneumonia is one of the most frequent and most severe medical complications in patients hospitalized in intensive care units. It develops mainly in association with invasive airway management and mechanical ventilation. It is an important factor affecting health care economy and often related to bacterial resistance. Understanding the etiology of pathogens and their potential resistance to antimicrobial agents has a major impact on both patients' morbidity and mortality and the economic aspect of their treatment. Pneumonia is diagnosed by assessing clinical signs and detecting etiologic agents. Clinical signs are assessed especially by finding fresh or progressive infiltrates on chest radiographs, together with at least two other signs of respiratory tract infection. From the epidemiological point of view, pneumonia may be either community-acquired (CAP) or hospital-acquired (HAP). CAP is defined by developing in the community outside health care facilities and, if the patient is hospitalized, clinical manifestations within 48 h of hospital admission. HAP may be characterized as pneumonia developing 48 h or more after admission to a health care facility or within 14 days after discharge. More precise classification according to the time of the onset of clinical signs distinguishes early-onset (from 2 to 4 days after admission) from late-onset (from day 5 after admission) HAP. The most common pathogens causing CAP are Streptococcus pneumoniae, Chlamydophila pneumoniae and Mycoplasma pneumoniae. HAP is mostly caused by endogenous bacterial strains, originating from primary microflora or secondary colonizing bacteria with a higher level of resistance in the early- and late-onset forms, respectively. This knowledge is used to select the proper therapy since the proportion of individual pathogens determines the strategy of initial antibiotic treatment. Adequate antibiotic therapy is an important factor influencing the effectiveness of therapy and, of course, the patient's survival. The prospective study aimed at identifying etiologic agents of pulmonary inflammation in patients with the most severe forms of respiratory insufficiency requiring mechanical ventilation. The objectives were to describe the prevalence of respiratory tract pathogens, to determine their susceptibility to a range of tested antibiotic agents, and to acquire information on the proportion of resistant strains in the population of these pathogens. The impact of adequate antibiotic therapy was assessed, with respect to patient mortality and morbidity rates.

Hypothesis. Most sever types of nosocomial bacterial pneumonias, required artificial lung ventilation are often exogenous. The infection source is transferred to patient´s airways from outsider during hospitalisation. The object of the research is bacterial agent direct recognition, its originality identification based on genome restrict fragment analysis.

Material and Methods. The group comprised patients hospitalized in the Intensive Care Departments of cooperating hospitals between 1 May 2013 and 30 April 2015 who developed signs of HAP. Also included are patients with positive findings in their tracheal secretion on admission to the department if transferred from another ward of the hospital. In intubated patients, secretion samples for microbiology culture tests are obtained by aspiration from the lower airway. Mortality is statistically analyzed by Fisher's exact test. The clinical signs of pneumonia are defined as the presence of newly developed or progressive infiltrates on chest radiographs plus at least two other signs of respiratory tract infection: temperature >38 °C, purulent sputum, leukocytosis >10x103/mm3 or leukopenia <4x103/mm3, signs of inflammation on auscultation, cough and/or respiratory insufficiency with oxygenation index≤300 mm Hg. Each sample is processed by semiquantitative method based on the four-quadrant streak technique using a calibrated loop. The etiologic agent is considered relevant if cultured in the tracheal secretion at a enough quantity. Tracheal secretion samples are processed by traditional microbiological methods. The microorganisms are identified by biochemical dentification tests, and automated systems. The yeasts are identified using commercial kit. If an identical culture, determined as the etiologic agent, is repeatedly isolated from multiple samples obtained from the same patient, only the first isolated culture is included in the study. Susceptibility to antibiotics is determined by the standard microdilution method. Adequate initial therapy is defined as administrative of at least one antibiotic (suitable for treating pneumonia) shown in vitro to be effective against the isolated causative agent.

Progress chart. The collection and processing of the patient´s microbiological samples at cooperatived clinic departments between 1 May 2013 and 30 April 2015 will be performed. The co-operative centers sent the samples to microbiological departments of their own hospitals and there the samples will processed and safed. Collected data will continuously to the central database be stored. The microbiological samples collection will finish 30 April 2015 and between 1 May 2015 and 31 december 2015 the data will be analysed and assessed. The processing of the data allows express conclusions and prepare proposals to event. hygienical arrangement changes.

Way of data acquiring. In intubated patients, secretion samples for microbiology culture tests were obtained by aspiration from the lower airway. The group comprise patients hospitalized in the Intensive Care Department of Hospitals, cooperated in study, between 1 May 2013 and 30April 2015 who developed signs of HAP. Also included are patients with positive findings in their tracheal secretion on admission to the department if transferred from another ward of the hospital. Predicted number of patients is 300 (400 - 500 positive isolates). Considerate number is estimated according the pilot study. Predicted number of patients in all cooperated centers is about 15 per month. There the data analysis will be made with statistic normality test Shapiro-Wilk and Mann-Whitney U test. Computer program SPSS version 15 to statistic assessment will be used.

Cooperation. The project is multicentric. There are cooperating Departments of Anesthesiology and Intensive Care Medicine in Olomouc, Brno, Hradec Kralove and Thomayer's Hospital Praha. The assessing of microbiological samples, collected from patients in this hospitals will be in microbiologic departments of this hospitals made.

Discussion. Given the incidence of 51 cases out of a total of 508 patients hospitalized in the Department of Anesthesiology and Intensive Care Medicine Olomouc, Czech Republic, in 2011, the prevalence (10%) was at the lower limit of the commonly reported range (9-24%). In agreement with the literature, most cases (86%) were late-onset HAP. Bacterial pathogens associated with the majority of deaths were strains of Klebsiella pneumoniae, Pseudomonas aeruginosa, Burgholderia cepacia komplex and Escherichia coli, more than 50% of which were multiresistant. In late-onset HAP, multiresistant strains accounted for as many as 58% of strains. In early onset HAP, the proportion of multiresistant strains could not been reliably assessed due to the small number of cases. The mortality rates in patients receiving adequate initial antibiotic therapy were 13% lower than in those treated with antibiotics to which isolated bacterial pathogens were later found to be resistant. According to Fiser's two-sided exact test, the resulting difference in mortality rates between the two studied groups is not significant (P=0.385), because of small set of data. Given the fact that despite adequate initial antibiotic therapy, the mortality rates were relatively high (9 out of 30 dead patients) and mortality is also likely to be influenced by the time of initiation of antibiotic therapy. In case of the mortality rates in patients with adequate therapy, our results (30%) are in agreement with those by Luna et al. who reported 38%. The same authors also found 91% mortality associated with inadequate therapy, a much higher rate than our results (43%). The difference, however, might be explained by a different epidemiological situation at bacterial resistance levels. HAP may be characterized as endogenous. Despite the high proportion of multiresistant strains, clonal spread was not confirmed, with the exception of Burgholderia cepacia komplex. Thus, secondary colonization of patient's microflora during hospitalization is likely.

ELIGIBILITY:
Inclusion Criteria:

* The clinical signs of pneumonia are defined as the presence of newly developed or progressive infiltrates on chest radiographs plus at least two other signs of respiratory tract infection: temperature >38 °C, purulent sputum, leukocytosis >10x103/mm3 or leukopenia <4x103/mm3, signs of inflammation on auscultation, cough and/or respiratory insufficiency with oxygenation index PaO2/FiO2 ≤300 mm Hg.

Exclusion Criteria:

* Pregnancy.
* The etiologic agent is considered relevant if cultured in the tracheal secretion at a quantity of >105 CFU/ml.
* Patients agreement absence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The group comprised patients hospitalized in the Intensive Care Departments of cooperating hospitals between 1 May 2013 and 30 April 2015 who developer signs of HAP.
Sampling Method: Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2013-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Mortality scale | 30 days
  Mortality scale YES/NO

SECONDARY OUTCOMES:
Initial empiric antibiotic therapy adequacy scale | 1 day
  Initial empiric antibiotic adequacy scale YES/NO